CLINICAL TRIAL: NCT02105181
Title: Temporary Placement of Fully Covered Self-expandable Metal Stents in Benign Biliary Strictures
Brief Title: Fully Covered Self-expandable Metal Stents (FCMS) in Benign Biliary Strictures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société Française d'Endoscopie Digestive (Other)
Responsible Party: Principal Investigator, Chaput Ulriikka, Dr Ulriikka Chaput, Société Française d'Endoscopie Digestive
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-A00197-44
Record Dates: First submitted 2014-04-02; First posted 2014-04-07 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Biliary Stricture
Keywords: benign biliary stricture; anastomotic biliary stricture after liver transplantation; chronic pancreatitis; biliary surgical procedure; fully covered metal stent
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fully covered metal stent (FCMS) (Other): There is one arm in the study : the intervention consists on placing a device which is a fully covered metal stent in the biliary tract of all patients
  Interventions: Device: Placement of a FCMS in the biliary tract of the patients

INTERVENTIONS:
Device: Placement of a FCMS in the biliary tract of the patients — During an ERCP procedure, a fully covered biliary metal stent (FCMS) is placed across a benign biliary stricture

SUMMARY:
Endoscopic treatment of benign biliary strictures can be challenging. Balloon dilation and/or plastic stent placement are currently the most popular techniques. Partially covered self-expandable metallic stents have also shown to be effective but can be difficult to remove. A novel fully covered metallic stent has recently been developed.

The aim of this study was to prospectively evaluate the placement of fully covered self-expandable metallic stents (FCSEMS) in this setting.

DETAILED DESCRIPTION:
After inclusion, an endoscopic procedure (ERCP) was performed in all patients in order to place a FCMS across the benign biliary stricture. The FCMS was left in place for 6 months and then extracted during a second ERCP procedure. An opacification was performed to assess the efficacy of stenting. Patients were followed up during one year after FCMS extraction.

ELIGIBILITY:
Inclusion Criteria:

* a history of liver transplantation, chronic pancreatitis or biliary surgery
* impairment of liver function tests such as elevated liver enzymes and/or cholestasis
* a biliary stricture associated with ductal dilation detected by US, CT or MRI, with a minimum distance of 2cm between the upper stricture's edge and the lower limit of the main biliary confluence or liver hilum .

Exclusion Criteria:

* an uncertainty about the benign nature of the stricture
* an intra-hepatic cholangitis and/ or a stricture extending beyond the hilum

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2007-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Initial success rate of temporary FCMS placement | 6 months
  Absence of biliary stricture or as an attenuated stricture on cholangiogram after removal of FCMS

SECONDARY OUTCOMES:
Final success | 18 months
  Absence of biliary stricture or the presence of an attenuated stricture and normal liver function tests at the end of follow up.
Stricture recurrence | 18 months
  Both clinically and ERCP-documented recurrence of stricture after an initial success.

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Prat, MD, PhD, Principal Investigator — Société Française d'Endoscopie Digestive
Locations (1):
- Hôpital Cochin, Paris, France